CLINICAL TRIAL: NCT05041556
Title: Strengthening the Evidence for Policy on the RTS,S/AS01 Malaria Vaccine: Assessment of Safety and Effectiveness Using Case-control Studies Embedded in the Malaria Vaccine Pilot Evaluation
Brief Title: Strengthening the Evidence for Policy on the RTS,S/AS01 Malaria Vaccine
Acronym: MVPE-CC
Status: Recruiting | Type: Observational
Sponsor: Kintampo Health Research Centre, Ghana (Other)
Collaborators: European Vaccine Initiative (Other); London School of Hygiene and Tropical Medicine (Other); African Research Collaboration for Health Limited (Unknown); Kenya Medical Research Institute (Other); University of Malawi (Other); PATH (Other)
Responsible Party: Sponsor
Other Study IDs: GHS-ERC 006/01/21
Record Dates: First submitted 2021-08-20; First posted 2021-09-13 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Malaria
Keywords: Malaria; Vaccines; Case-control; Safety; Mortality
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Case-control study of clinical outcomes: These are children who live in RTS,S implementation areas aged less than 5 years and who were eligible to have received RTS,S based on their date or birth and age, will be eligible to be recruited into the study. Cases will be recruited in sentinel hospitals of the ongoing malaria Vaccine Pilot Evaluation (MVPE). Control for a case will be a child who lives outside a 100-metre radius from the case, matched on date of birth (+/- 1 month of date of birth of the case)
  Interventions: Other: Case-control study of clinical outcomes
- Case-control study of mortality outcome: These will be children who died of any cause excluding accidents or trauma, who are eligible to have received the RTS,S vaccine based on their date of birth and age. Cases will be recruited from the community-based mortality surveillance of MVPE. Control for a mortality case will be a live child who lives outside a 100 metre radius from the case with date of birth +/- 1 month of the date of birth of the case who are eligible to have received the RTS,S vaccine.
  Interventions: Other: Case-control study of mortality outcome

INTERVENTIONS:
Other: Case-control study of clinical outcomes — A case-control questionnaire will be administered at the home of cases and controls
  Groups: Case-control study of clinical outcomes
Other: Case-control study of mortality outcome — A case-control questionnaire will be administered at the home of cases and controls
  Groups: Case-control study of mortality outcome

SUMMARY:
The ongoing Malaria Vaccine Pilot Evaluation (MVPE) is being conducted in Ghana, Malawi and Kenya through community and sentinel hospital surveillance systems and a series of household surveys (to measure vaccine coverage). The Malaria Vaccine Pilot Evaluation-Case Control (MVPE-CC) registered here as observational study is embedded within MVPE comprising case-control studies of clinical and mortality outcomes. Each case will require four controls, and caregiver informed consent will be required prior to study activities.

These observational case control studies will measure as complementary information to what is being collected through MVPE:

1. Safety among children who received the malaria vaccine, with focus on cerebral malaria, meningitis and severe malaria
2. The impact of the malaria vaccine on all-cause mortality for boys and girls, AND
3. Promote use of case-control approaches by Expanded Programmes on Immunization (EPI) and malaria control programmes.

DETAILED DESCRIPTION:
Strengthening the evidence for policy on the RTS,S/AS01 malaria vaccine: assessment of safety and effectiveness using case-control studies embedded in the Malaria Vaccine Pilot Evaluation (MVPE). This project will support the embedding of case-control studies into the ongoing evaluation component of the RTS,S malaria vaccine pilot implementation programme (MVIP) in Ghana, Kenya, and Malawi. The evaluation data are being collected through a series of household surveys, and sentinel hospital and community mortality surveillance build on routine systems.

The case-control studies will run for a period of 45 months in the three countries (Ghana, Kenya, Malawi). The primary objectives of the case-control studies focus on safety, impact and capacity building. There will be no defined number of cases per country. Data for the case-control studies will be collected using two-pronged approach.

CASE-CONTROL STUDY OF CLINICAL OUTCOMES.

For each case, 4 controls will be recruited.

Children living in the study area of the ongoing MVPE and recruited from the catchment areas of the sentinel hospital of the MVPE will be recruited. Children aged 6 months - 59 months will be recruited into the study. All eligible cases identified from the MVPE sentinel hospital surveillance systems will be recruited. Data needed on cases already being collected as part of the MVPE sentinel surveillance will be updated following consent. Eligible cases will be approached for consent for the case-control component and to ascertain their residence and collect additional data. Neighbourhood controls will be recruited by canvassing homes in a predetermined pattern from the case's home until four eligible controls are identified and interviewed. Research officers will identify and consent controls. Similar information will be collected as for the cases. A total of 46 meningitis cases and 184 controls, and 930 severe malaria cases and 3720 controls will contribute to the clinical case-control endpoints across the three countries. This is expected to provide 90% power to detect a 10 to 5-fold increase in incidence of meningitis in vaccine recipients. The updated power calculations indicate about 600 severe malaria cases is needed to detect the 40% benefit that was seen in the phase 3 trial. And 330 severe malaria cases eligible to have received 3 doses (and not yet eligible for dose 4) are needed for 80% power to detect a 30% reduction in incidence. A total of 180 cases of cerebral malaria and 720 controls are expected to be recruited to provide 90% power to detect a 2-fold increase in incidence of cerebral malaria in children who received 3 doses of RTSS/AS01

CASE-CONTROL STUDY OF MORTALITY OUTCOMES.

For each case, 4 controls will be recruited.

As part of the MVPE, data is already captured on all children aged 1 - 59 months who live in an MVIP area and die by verbal autopsy teams at the child's home. Data already collected within the context of the MVPE will be merged to the case-control dataset using the child's unique identifier, rather than duplicated. For the mortality case-control outcomes, verbal autopsy teams will identify eligible deaths at the time of the verbal autopsy. Written, or witnessed and thumb-printed, informed consent will be obtained from each child's carer before data are included in the case-control dataset. Data may be captured retrospectively once the informed consent form is signed or thumb-printed.

Four controls will be selected per case, and matched based on their location and their age (within 30 days of the case's date of birth). To avoid selection bias, research officers will canvass up to several homes in a predetermined pattern from the case's home until four controls are identified and interviewed. All eligible controls will be approached for consent. The same information will be collected for controls as for the cases. A total of 1000 mortality cases and 4000 controls will contribute to the clinical case-control endpoints. This is expected to provide 90% power to detect a 2-fold difference between girls and boys.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate in study evidenced by written informed consent provided by an adult caregiver
* Resident in an RTS,S/AS01 implementation area within the catchment area of MVPE sentinel hospitals
* Eligible, based on date of birth and age, to have received RTSS/AS01
* Meets the case or control definitions above.

Exclusion Criteria:

* Caregiver not willing to provide consent

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population will comprise children aged 6-59 months who live in RTS,S implementation areas in Ghana, Kenya and Malawi and who were eligible to have received RTS,S based on their date or birth and age
Sampling Method: Non-Probability Sample
Enrollment: 9280 (Estimated)
Dates: Start 2021-10-18 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of children admitted with a diagnosis of probable and confirmed meningitis | Through study completion, an average of 1 year
  Number of children with probable and confirmed meningitis. A case of meningitis will include probable or confirmed meningitis, defined as a child eligible to have received the RTS,S vaccine and admitted with clinical signs of meningitis, CSF that is turbid, cloudy or purulent or with CSF leukocyte count >10 cells/mm3, or with a pathogen isolated at the central reference laboratory from CSF . A control to a meningitis case is defined as a child who lives outside a 100 metre radius from the case with date of birth within +/- 1 month of date of birth of the case, recruited concurrently with the case
Number of children admitted with a diagnosis of severe malaria | Through study completion, an average of 1 year
  Number of children admitted with a diagnosis of severe malaria. A case of severe malaria is defined as a child who was eligible to have received RTS,S and diagnosed as severe malaria based on the presence of Plasmodium falciparum parasitaemia detected by microscopy or rapid diagnostic test, with impaired consciousness, convulsions, respiratory distress, severe malarial anaemia (hemoglobin level < 8g/dL or requiring blood transfusion for anaemia) or cerebral malaria [ P. falciparum parasitaemia with impaired consciousness (Glasgow coma score <11 (children 2 years of age and above) or a Blantyre coma score <3 in children under 2 years or assessed as P or U on AVPU score) with a clinical diagnosis of cerebral malaria and CSF findings not consistent with meningitis]. A control for a severe malaria case will be defined as a child who lives outside a 100 metre radius from the case, matched on date of birth (+/- 1 month of date of birth of the case
The number of deaths of any cause | Through study completion, an average of 1 year
  The number of deaths of any cause. Cases will be children who died, of any cause excluding accidents or trauma, who are eligible to have received the RTS,S vaccine based on their date of birth and age. A control to a mortality case will be defined as a live child who lives outside a 100 metre radius from the case with date of birth +/- 1 month of the date of birth of the case who are eligible to have received the RTS,S vaccine.
Number of deaths in children by gender | Through study completion, an average of 1 year
  Number of deaths in children stratified by gender in children aged 6-59 months

SECONDARY OUTCOMES:
Number of children with a diagnosis of severe malaria in relation to the 4th dose of RTS,S | Through study completion, an average of 1 year
  Hospital admissions with malaria which meet WHO criteria for a diagnosis of severe malaria
Number of children with a diagnosis of cerebral malaria in relation to the 4th dose of RTS,S | Through study completion, an average of 1 year
  Hospital admissions with malaria which meet WHO criteria for a diagnosis of cerebral malaria
Number of deaths of any cause in relation to the 4th dose of RTS,S | Through study completion, an average of 1 year
  Number of deaths of any cause in relation to the 4th dose of RTS,S among children aged 6-59 months.
Number of deaths among girls in relation to the 4th dose of RTS,S | Through study completion, an average of 1 year
  Number of deaths in children stratified by gender in relation to the 4th dose of RTS,S among children aged 1-59 months

CONTACTS AND LOCATIONS:
Overall Officials: Kwaku Poku Asante, PhD, Principal Investigator — Kintampo Health Research Centre, Ghana; Don Mathanga, PhD, Principal Investigator — College of Medicine, University of Malawi, Malawi; Samuel Akech, PhD, Principal Investigator — African Research Collaboration for Health Limited, Kenya; Simon Kariuki, PhD, Principal Investigator — Kenya Medical Research Institute
Locations (4):
- Kintampo Health Research Centre, Kintampo, Ghana
- Kenya (2):
  - African Research Collaboration for Health Limited, Nairobi
  - Kenya Medical Research Institute (KEMRI), Nairobi
- College of Medicine, University of Malawi, Blantyre, Malawi